CLINICAL TRIAL: NCT04866433
Title: The Effect of Real-time Binaural Sound on Sedation Using Dexmedetomidine During Spinal Anesthesia: a Randomized, Placebo-controlled Trial
Brief Title: The Effect of Real-time Binaural Sound on Sedation Using Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2101-185-1193
Record Dates: First submitted 2021-04-19; First posted 2021-04-29 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Sedative Adverse Reaction
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Binaural group (Experimental): Play realtime binaural sound applied music through headphones
  Interventions: Procedure: Real-time binaural sound
- Audio group (Active Comparator): Play music through headphones.
  Interventions: Procedure: Music
- Control group (Sham Comparator): Wear headphones that do not produce sound.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Real-time binaural sound — Play music with a frequency difference (real-time binaural sound) in each ear through headphones during sedation.
  Arms: Binaural group
Procedure: Music — Play the same music in both ears through headphones during sedation
  Arms: Audio group
Procedure: Control — Just wear headphones during sedation
  Arms: Control group

SUMMARY:
The aim of the study is to evaluate whether real-time binaural sound affects the dose of dexmedetomidine in patients undergoing sedation with dexmedetomidine after spinal anesthesia.

DETAILED DESCRIPTION:
Patients undergoing sedation with dexmedetomidine after spinal anesthesia are randomly assigned to binaural group, audio group, and control group. After spinal anesthesia, SedLine continuous monitoring is started. Real-time binaural sound applied music is played to the binaural group, normal music is played to the audio group, and headphones with no sound are applied to the control group. Observer's Assessment of Alertness/Sedation Scale (OAAS) and Patient State Index (PSi) are checked every minute after loading of dexmedetomidine at the rate of 1 μg/kg for 10 minutes (6 μg/kg/hr). Loading is stopped when the OAAS score is 3 or less. Then, dexmedetomidine is continuously infused at a rate of 0.6 μg/kg/hr, and OAAS is evaluated every 30 minutes. The infusion rate is lowered (-0.1 μg/kg/hr) if OAAS is lower than 3, and increased (+0.1 μg/kg/hr) if OAAS is higher than 3. The continuous infusion rate should not exceed 1 μg/kg/hr. The total dexmedetomidine dose corrected by the patient's predicted body weight and infusion time (μg/kg/hr) was compared between groups. In addition, the loading dose (μg/kg) and continuous infusion dose (μg/kg/hr), additional sedative use, blood pressure, heart rate, ECG changes, respiratory depression, and oxygen saturation were observed. The patient's satisfaction is evaluated after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing sedation with dexmedetomidine during spinal anesthesia for surgery with an estimated time of 90 minutes or longer

Exclusion Criteria:

* ASA physical status classification 3-4
* Patients with hearing loss or using hearing aids
* Patients who received narcotic analgesics or sedative drugs within 1 week
* Patients with alcohol dependence or drug dependence
* Patients with drug hypersensitivity to dexmedetomidine
* Patients with arrhythmia, cardiovascular disease, decreased cardiac function and decreased cardiac output
* Patients who are judged to be difficult to use sedative drugs due to severe respiratory disease
* Patients with liver failure
* Patients with kidney failure or on dialysis
* Patients judged to be unsuitable for the clinical trial by the researchers
* Patients whose actual operation time is less than 30 minutes

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Dexmedetomidine loading dose injected until OAAS reaches 3 or less (μg/kg) | Intraoperative (During sedation for surgery)
  Dexmedetomidine loading dose injected until OAAS reaches 3 or less (μg/kg)

SECONDARY OUTCOMES:
Observer's Assessment of Alertness/Sedation Scale (0~5) | During sedation for surgery and at post anesthesia care unit (PACU)
  Observer's Assessment of Alertness/Sedation Scale (0, does not respond to painful trapezius squeeze; 1, responds only after painful trapezius squeeze; 2, responds only after mild prodding or shaking; 3, responds only after name is called loudly, repeatedly, or both; 4, responds lethargically to name spoken in normal tone; 5, responds readily to name spoken in normal tone)
Patient State Index (PSi) | Intraoperative (During sedation for surgery)
  Patient State Index (PSi) acquired through the Sedline Sedation monitor (Sedline, Massimo, USA)
Dexmedetomidine continuous infusion dose | Intraoperative (During sedation for surgery)
  Total amount of dexmedetomidine infused from the end of dexmedetomidine loading to the start of suturing the surgical site
Number of patients requiring additional sedatives | Intraoperative (During sedation for surgery)
  Number of patients requiring additional sedatives
Adverse event | Intraoperative (During sedation for surgery)
  Incidence of hypotension, hypertension, bradycardia, ECG change, need of vasopressors, respiratory suppression, desaturation
Patient satisfaction | Intraoperative (At the time of leaving the operating room)
  Patient's satisfaction with intraoperative sedation Score from 0 to 10) with intraoperative sedation measured at the time of leaving the operating room (0~10)
Postanesthesia recovery score (0~10) | At the postanesthesia recovery room
  Postanesthesia recovery score (0~10, higher scores mean better recovery)
Postoperative delirium | From the end of the surgery to the hospital discharge, an average of 1 week
  Incidence of postoperative delirium

OTHER OUTCOMES:
EEG power in delta band | During sedation for surgery
  EEG power in delta band (0.3~4Hz) acquired through the Sedline Sedation monitor (Sedline, Massimo, USA)
EEG power in theta band | During sedation for surgery
  EEG power in theta band (4~8Hz) acquired through the Sedline Sedation monitor (Sedline, Massimo, USA)
EEG power in alpha band | During sedation for surgery
  EEG power in alpha band (8~13Hz) acquired through the Sedline Sedation monitor (Sedline, Massimo, USA)
EEG power in beta band | During sedation for surgery
  EEG power in beta band (13~30Hz) acquired through the Sedline Sedation monitor (Sedline, Massimo, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Bae J, Yoo S, Kim H, Kim Y, Kim JT, Lim YJ, Kim HS. Effect of real-time binaural music on sedation with dexmedetomidine during spinal anesthesia: A triple-arm, assessor-blind, randomized controlled trial. J Clin Anesth. 2023 Feb;84:110997. doi: 10.1016/j.jclinane.2022.110997. Epub 2022 Nov 10. PMID 36371942